CLINICAL TRIAL: NCT07296003
Title: A Longitudinal Observational Study of Early Spontaneous Motor Activity, Postural Control, and Motor Optimality Score (MOS-R) as Predictors of Psychomotor, Cognitive, and Sensory Development at 18 and 36 Months in Preterm and Term Infants, With Consideration of Early Therapeutic Intervention
Brief Title: Motor Development and Early Predictors of Psychomotor Outcomes in Preterm and Term Infants Assessed by MOS-R and Caregiver Questionnaire at 18 and 36 Months
Status: Recruiting | Type: Observational
Sponsor: Masaryk University (Other)
Responsible Party: Sponsor
Other Study IDs: 707/19.4.2024
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Neurodevelopmental Disorders; Motor Skills Disorders; Infant, Premature Development; Infant, Term Development; Postural Balance
Keywords: General Movements Assessment; Motor Optimality Score Revised; Postural Control; Full-Term Infants; Preterm Infants; Neurodevelopmental Outcomes
MeSH Terms: conditions — Neurodevelopmental Disorders; Motor Skills Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm Infants Cohort: Infants born moderately or late preterm (32-36 weeks gestation) who completed standardized video-based assessment of early spontaneous movements in infancy. Within this cohort, infants will be further stratified according to the quality of early spontaneous movements as evaluated by the Motor Optimality Score - Revised (MOS-R), distinguishing between typical movement quality and reduced or atypical movement quality. Among infants showing reduced or atypical movement quality, naturally occurring differences in early physiotherapy exposure will also be described. These characteristics serve as analytic stratification factors and do not define additional study groups.
  Interventions: Other: Vojta method
- Full-Term Infants: Infants born at or after 37 weeks of gestation who completed the same standardized early assessment of spontaneous movements. As in the preterm cohort, infants will be stratified based on the quality of early spontaneous movements assessed using the Motor Optimality Score - Revised (MOS-R), distinguishing between typical and reduced or atypical movement quality. For infants with reduced/atypical movement quality, differences in early physiotherapy exposure may also be explored. These variables function as stratification factors for analysis and are not defined as separate study cohorts.
  Interventions: Other: Vojta method

INTERVENTIONS:
Other: Vojta method — Vojta method, also known as reflex locomotion, was offered to infants who demonstrated atypical or reduced quality of early spontaneous motor behavior during clinical evaluation. The method uses specific pressure stimulation zones to activate innate locomotor patterns aimed at improving postural control, axial stability, and motor coordination. In this study, Vojta therapy was not assigned by the research protocol but initiated by caregivers following clinical recommendation. Therefore, exposure to Vojta method represents a naturally occurring, non-randomized behavioral intervention and is analyzed only for exploratory purposes.

SUMMARY:
This study examines how early motor behavior in infants relates to their later psychomotor development. Researchers will observe both preterm and full-term infants during the first months of life, using video-based assessments to evaluate spontaneous movements and early postural control. These early motor patterns will be scored with the Motor Optimality Score - Revised (MOS-R).

When the children reach 18 and 36 months of age, their development in areas such as motor skills, communication, sensory processing, and social behavior will be evaluated through a caregiver-completed questionnaire.

The purpose of the study is to determine whether early motor quality can predict later developmental outcomes, whether preterm and full-term infants with similar motor scores develop differently, and whether early therapy may improve outcomes for infants with low MOS-R results.

DETAILED DESCRIPTION:
This study uses a combined retrospective-prospective observational design. The retrospective component includes previously recorded video assessments of spontaneous motor behavior and postural control collected during routine clinical examinations in both preterm infants and a comparison group of full-term infants. These recordings were originally obtained as part of standard care in the neonatal unit and physiotherapy outpatient clinic and were subsequently anonymized for research purposes. Early motor quality was evaluated using standardized scoring procedures, including the Motor Optimality Score - Revised (MOS-R) and detailed general movement assessment.

The prospective component is used to complete developmental follow-up. Caregivers are contacted when the child reaches 18 and 36 months of age and are asked to complete a validated questionnaire assessing domains such as motor development, communication, sensory processing, and socio-emotional functioning. By integrating retrospective motor assessments with prospective developmental outcomes, the study enables a rigorous analysis of the predictive relationship between early motor patterns and later psychomotor development.

A combined design is necessary because high-quality video recordings of early motor behavior cannot be reproduced once the infant has aged, and the early spontaneous movement repertoire represents a unique neurodevelopmental window. The retrospective use of existing recordings reduces participant burden and allows comparison between preterm infants and full-term infants who underwent the same standardized motor assessment. The prospective follow-up ensures that developmental outcomes are measured consistently and with sufficient temporal precision. Overall, this design increases feasibility, minimizes risk, and provides a robust framework for evaluating early markers of developmental trajectories.

ELIGIBILITY:
Inclusion Criteria:

* The child was born either preterm or full-term. Both groups are included in the study.
* The child completed a video recording of early movements during routine check-ups in the first months of life.
* The parents or legal guardians agree to participate and give informed consent.
* The child will be available for follow-up at around 18-36 months of age, when parents will complete a developmental questionnaire.

Exclusion Criteria:

* There is no usable video recording of the child's early spontaneous movements from the neonatal or early infant period.
* The child has a diagnosed medical condition that makes movement assessment impossible (for example, severe congenital anomalies or conditions preventing typical movement).
* Parents do not wish to participate or withdraw their consent.
* The child is not available for follow-up, meaning that the developmental questionnaire at 18-36 months cannot be completed.

Max Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants in this study are infants who were seen for routine clinical follow-up in the Neonatal Unit and the physiotherapy outpatient clinic at Pardubice Regional Hospital and cooperating rehabilitation centers. During their early visits, these infants had video recordings made of their spontaneous movements as part of standard clinical care. Both preterm and full-term infants are included. When the children reach approximately 18-36 months of age, their parents or legal guardians are invited to complete a developmental questionnaire as part of the study's follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2026-07-28 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Association Between the Quality of Early Spontaneous Movements and Developmental Outcomes at 18 and at 36 months | april 2024 - july 2027
  The quality of early spontaneous movements will be evaluated using standardized observational assessment in infancy. Developmental outcomes at 18 and 36 months will be compared between infants displaying typical movement quality and those showing reduced or atypical movement quality. This analysis aims to determine whether early differences in spontaneous motor behavior are associated with variations in later developmental functioning.

SECONDARY OUTCOMES:
Correlation Between MOS-R and Specific Developmental Sub-Domains (Motor vs. Non-Motor) | april 2024 - july 2027
  Assessment of the relationship between early MOS-R scores and specific sub-scales of the caregiver questionnaire at both 18 and 36 months. The analysis will distinguish between Gross/Fine Motor scores versus Communication and Social-Emotional scores. The aim is to evaluate whether early motor optimality is a stronger predictor of later motor skills compared to cognitive/language skills.

OTHER OUTCOMES:
Predictive Validity of MOS-R in Preterm vs. Full-Term Cohorts | april 2024 - july 2027
  Comparison of the association strength between MOS-R and later developmental outcomes in the Preterm cohort (born <37 weeks) versus the Full-Term cohort. This measure investigates whether the predictive value of early motor assessment differs based on gestational age at birth.
Developmental Outcomes in Infants With Atypical Early Movement Quality Who Did or Did Not Receive Early Therapy | april 2024 - july 2027
  Among infants displaying atypical or reduced quality of early spontaneous movements, developmental outcomes at 18 and 36 months will be compared based on whether families chose to initiate early physiotherapy. Because group assignment is based on parental decision-making and not randomization, this outcome is exploratory and may be influenced by indication bias.

CONTACTS AND LOCATIONS:
Locations (2):
- Czechia (2):
  - Nemocnice Pardubického kraje, a.s., Pardubice, Czechia
  - Lentilka - integrated kindergarden and rehabilitation center, Pardubice, Česká Republika

IPD SHARING:
Plan to Share IPD: No